CLINICAL TRIAL: NCT04797546
Title: Impact of Adductor Canal Block, Compared to Patient Controlled Analgesia, in the Surgical Stress Response of Patients Programmed for Traumatic Anterior Cruciate Ligament Repair
Brief Title: Adductor Canal Block Versus Patient Controlled Analgesia, in the Surgical Stress Response for Anterior Cruciate Ligament Repair
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-128
Record Dates: First submitted 2016-09-12; First posted 2021-03-15 (Actual); Last update posted 2021-03-15 (Actual); Status verified 2016-09

CONDITIONS: Anesthesia; Stress, Physiological; Surgery
MeSH Terms: interventions — Analgesia, Patient-Controlled

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Adductor Canal Block (Experimental): With mild sedation, a continous bupivacaine 0.1% infusion catheter is placed in the adductor canal. Afterwards, patients are placed under General Anesthesia, and surgery starts. Preoperative, 2 hours and 24 hours stress biomarkers and analgesic quality will be measured.
  Interventions: Procedure: Adductor Canal Block
- Patient Controlled Morphine Analgesia (Active Comparator): Patients are placed under General Anesthesia, and after surgery, a Morphine patient controlled analgesia delivery system is installed. Preoperative, 2 hours and 24 hours stress biomarkers and analgesic quality will be measured.
  Interventions: Device: Morphine Patient Controlled Analgesia

INTERVENTIONS:
Procedure: Adductor Canal Block — Continous peripheral nerve block
  Arms: Adductor Canal Block
Device: Morphine Patient Controlled Analgesia — Morphine Patient Controlled Analgesia Delivery System
  Other Names: Patient Controlled Analgesia
  Arms: Patient Controlled Morphine Analgesia

SUMMARY:
To evaluate the surgical stress response in anterior cruciate ligament repair with an adductor canal block versus patient controlled endovenous analgesia.

DETAILED DESCRIPTION:
Preoperative, 2 hours and 24 hours stress biomarkers will be evaluated in two groups of patients, continous adductor canal block and morphine patient controlled endovenous analgesia.

ELIGIBILITY:
Inclusion Criteria:

* Male,
* 18-65 years,
* traumatic Anterior Cruciate Ligament tear, scheduled for elective arthroscopic repair with Semitendinous-Gracillis technique at first time in the morning, with full articular range,
* no other traumatologic lesions.

Exclusion Criteria:

* denied consent to participate,
* chronic steroids user,
* diabetes type 1 or 2,
* insulin resistance,
* concurrent infectious disease,
* cognitive failure, coagulopathy,
* allergy to study drugs,
* surgery scheduled in the afternoon

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-09; Primary Completion 2018-05 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
Change of Blood Cortisol from baseline to 24 hours | 24 hours
  Blood Cortisol will be evaluated preoperatively, 2 hours and 24 hours postoperatively.

SECONDARY OUTCOMES:
Change of C Reactive Protein from baseline to 24 hours | 24 hours
  C Reactive Protein will be evaluated preoperatively, 2 hours and 24 hours postoperatively.
Change of Glycemia from baseline to 24 hours | 24 hours
  Glycemia will be evaluated preoperatively, 2 hours and 24 hours postoperatively.

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Altermatt, MD, Principal Investigator — PUC
Locations (1):
- Pontificia Universidad Católica de Chile, Santiago, Chile

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Desborough JP. The stress response to trauma and surgery. Br J Anaesth. 2000 Jul;85(1):109-17. doi: 10.1093/bja/85.1.109. No abstract available. PMID 10927999
- [Background] Weissman C. The metabolic response to stress: an overview and update. Anesthesiology. 1990 Aug;73(2):308-27. doi: 10.1097/00000542-199008000-00020. PMID 2200312
- [Background] Richardson J, Sabanathan S, Jones J, Shah RD, Cheema S, Mearns AJ. A prospective, randomized comparison of preoperative and continuous balanced epidural or paravertebral bupivacaine on post-thoracotomy pain, pulmonary function and stress responses. Br J Anaesth. 1999 Sep;83(3):387-92. doi: 10.1093/bja/83.3.387. PMID 10655907
- [Background] Hong JY, Yang SC, Yi J, Kil HK. Epidural ropivacaine and sufentanil and the perioperative stress response after a radical retropubic prostatectomy. Acta Anaesthesiol Scand. 2011 Mar;55(3):282-9. doi: 10.1111/j.1399-6576.2010.02360.x. Epub 2010 Nov 25. PMID 21108620
- [Background] Ahlers O, Nachtigall I, Lenze J, Goldmann A, Schulte E, Hohne C, Fritz G, Keh D. Intraoperative thoracic epidural anaesthesia attenuates stress-induced immunosuppression in patients undergoing major abdominal surgery. Br J Anaesth. 2008 Dec;101(6):781-7. doi: 10.1093/bja/aen287. Epub 2008 Oct 15. PMID 18922851
- [Background] Fant F, Tina E, Sandblom D, Andersson SO, Magnuson A, Hultgren-Hornkvist E, Axelsson K, Gupta A. Thoracic epidural analgesia inhibits the neuro-hormonal but not the acute inflammatory stress response after radical retropubic prostatectomy. Br J Anaesth. 2013 May;110(5):747-57. doi: 10.1093/bja/aes491. Epub 2013 Jan 7. PMID 23295713
- [Background] Bagry H, de la Cuadra Fontaine JC, Asenjo JF, Bracco D, Carli F. Effect of a continuous peripheral nerve block on the inflammatory response in knee arthroplasty. Reg Anesth Pain Med. 2008 Jan-Feb;33(1):17-23. doi: 10.1016/j.rapm.2007.06.398. PMID 18155052
- [Background] Fowler SJ, Symons J, Sabato S, Myles PS. Epidural analgesia compared with peripheral nerve blockade after major knee surgery: a systematic review and meta-analysis of randomized trials. Br J Anaesth. 2008 Feb;100(2):154-64. doi: 10.1093/bja/aem373. PMID 18211990
- [Background] Martin F, Martinez V, Mazoit JX, Bouhassira D, Cherif K, Gentili ME, Piriou P, Chauvin M, Fletcher D. Antiinflammatory effect of peripheral nerve blocks after knee surgery: clinical and biologic evaluation. Anesthesiology. 2008 Sep;109(3):484-90. doi: 10.1097/ALN.0b013e318182c2a1. PMID 18719447
- [Background] Cuellar VG, Cuellar JM, Golish SR, Yeomans DC, Scuderi GJ. Cytokine profiling in acute anterior cruciate ligament injury. Arthroscopy. 2010 Oct;26(10):1296-301. doi: 10.1016/j.arthro.2010.02.011. PMID 20887928
- [Background] Sharma A, Aoun P, Wigham J, Weist S, Veldhuis JD. Gender determines ACTH recovery from hypercortisolemia in healthy older humans. Metabolism. 2013 Dec;62(12):1819-29. doi: 10.1016/j.metabol.2013.08.014. Epub 2013 Sep 25. PMID 24074810